CLINICAL TRIAL: NCT04690010
Title: A Randomized Controlled Trial of Ambulatory Versus Inpatient Percutaneous Nephrolithotomy
Brief Title: Ambulatory Versus Inpatient Percutaneous Nephrolithotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-33137
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulatory tubeless PCNL (Active Comparator): Patients will be discharged home on the same day as surgery. No nephrostomy tube will be placed (tubeless).
  Interventions: Procedure: Ambulatory tubeless PCNL
- Inpatient PCNL with nephrostomy tube (Active Comparator): Patients will be admitted to hospital for 1-3 days with a nephrostomy tube placed at the time of surgery that will then be removed prior to discharge.
  Interventions: Procedure: Inpatient PCNL with nephrostomy tube

INTERVENTIONS:
Procedure: Ambulatory tubeless PCNL — Patients will be discharged the same day of surgery. No nephrostomy tube will be left in place. A ureteral stent on a string may be left for up to 5 days.
  Arms: Ambulatory tubeless PCNL
Procedure: Inpatient PCNL with nephrostomy tube — Patients will be admitted to hospital for 1-3 days. A nephrostomy tube will be placed at the time of surgery that will be removed prior to discharge.
  Arms: Inpatient PCNL with nephrostomy tube

SUMMARY:
The goal of the study is to determine if ambulatory tubeless PCNL is safe and effective compared to inpatient PCNL with a nephrostomy tube.

DETAILED DESCRIPTION:
One in eight human beings will develop kidney stones during their lifetime. Of these, roughly 20% require surgery. Percutaneous nephrolithotomy (PCNL) is the standard minimally invasive surgical procedure for removal of large kidney stones. In the standard PCNL technique, a drainage tube connecting the kidney to a bag on the outside of the body (nephrostomy tube) is left in place after surgery. Patients are admitted to hospital for one to two days for observation at which time the nephrostomy tube is removed before discharge. The presence of the nephrostomy tube is associated with pain, increased use of opioids, and slower recovery after surgery.

Ambulatory PCNL has been proposed as a way to potentially speed recovery, reduce pain, decrease time in hospital, and decrease cost. Initial studies of ambulatory tubeless PCNL have shown favourable results. However, these studies were performed in a small subset of healthy patients with favourable stones that do not represent the majority of patients who undergo PCNL. In this technique, patients are discharged home the same day as surgery usually with a small drainage tube on the inside of the body called a stent that is removed 1-2 weeks later and no nephrostomy tube (tubeless). The stent itself can be painful and may require a second procedure for removal. There is increasing evidence for the safety of totally tubeless PCNL (in which no nephrostomy tube or ureteric stent is placed) or placement of a stent on a string for a short period of time. Given that current recommendations for stone management in the times of COVID-19 include minimizing use of stents, the investigators believe it is an optimal time to evaluate safety and efficacy of using a minimal stenting technique (either no stent at all or stent on string) in ambulatory PCNL patients.

The goal of the study is to determine if ambulatory tubeless PCNL is safe and effective compared to inpatient PCNL with a nephrostomy tube in a more representative patient population including obese patients, patients with moderate medical comorbidities, and patients with large kidney stones. A secondary aim is to determine if a minimal stent technique (stent on a string for 5 days or less or no stent) is safe and effective as an exit strategy in ambulatory PCNL patients. The study hypothesis is that ambulatory tubeless PCNL will have similar complication and stone free rates as inpatient PCNL with benefits over inpatient PCNL including improved patient quality of life, decreased use of opioid pain medications, shortened hospital admission, faster return to work, and lower cost.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for PCNL who agree to be included in the study
* Age 18 years or more
* Absence of renal anatomic abnormalities
* Patients undergoing bilateral procedures or those with pre-operative indwelling ureteral stents or nephrostomy tubes will be included

Exclusion Criteria:

Pre-operative:

* Age <18
* Pregnancy
* Positive urine culture within 3 weeks
* Bleeding disorder
* Presence of renal anatomic abnormalities
* Solitary kidney
* Need for admission based on comorbidities determined by anesthesiologist

Intra-operative:

* Significant ureteral or pelvicalyceal injury
* Significant intraoperative hemorrhage

Post-operative:

* Temperature >100.4 Fahrenheit
* Hemodynamic instability (defined as 2 of 3: heart rate >90 beats per minute, respiratory rate >20 breaths per minute, systolic blood pressure <90mmHg, or drop in systolic blood pressure >40mmHg)
* Hemoglobin drop of > 3 g/dL compared to pre-operative bloodwork
* Transfusion of blood products
* Pneumothorax or hemothorax on chest X ray
* Uncontrolled nausea, vomiting, or pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-01-08 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Total number of complications | 4 weeks after surgery
  Any of: Emergency department visits related to procedure, unplanned provider visits, re-admission related to the procedure, blood transfusion, and need for secondary procedures. Patients with an emergency department or provider visit leading to re-admission will be classified once in the primary outcome as re-admission.

SECONDARY OUTCOMES:
Stone free status | 4 weeks after surgery
  Stone free status will be defined as no residual stones with maximum diameter >3 mm on low dose non-contrast CT scan at 4 weeks post-surgery.
Change in Wisconsin Stone Quality of Life Questionnaire by 10 points or more from baseline to 4 weeks after surgery. | This will be completed at the initial visit (baseline) and at the follow-up visit 4 weeks later.
  The Wisconsin Stone Quality of Life Questionnaire is a validated, disease specific quality-of-life instrument that has been used in the acute, chronic, and post-operative setting and is currently the most commonly used questionnaire for kidney stone disease.The survey is a 28-item instrument with a 5-point Likert scale for each item. There is a total of 140 points, and a difference of 10 points is considered clinically significant.
Cumulative opiate morphine equivalent dosing | 4 weeks after surgery
  This will be the calculated as the morphine equivalent dosage of all opioid medications taken by patients from time of surgery to follow-up at 4 weeks above their baseline opioid needs.
Return to work | 4 weeks after surgery
  Mean time to return to work (in days) and percent who have returned to work at 1 week will be determined at the time of the 4-week follow-up visit.
Time in hospital | 1 week after surgery
  Duration spent in hospital (in hours) will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No